CLINICAL TRIAL: NCT03662438
Title: HOPE (Home-based Oxygen [Portable] and Exercise) - Improving Mobility in Patients on Long Term Oxygen Therapy: a Home-based Physiotherapy Programme With Novel Ambulatory Oxygen Device.
Brief Title: HOPE (Home-based Oxygen [Portable] and Exercise) for Patients on Long Term Oxygen Therapy (LTOT)
Acronym: HOPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Singhealth Foundation (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE Study; SHF/HSRHO013/2017 (Other Grant/Funding Number: Singhealth Foundation)
Record Dates: First submitted 2018-08-29; First posted 2018-09-07 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Exercise Therapy; Physical Activity; Respiratory Failure; Oxygen Inhalation Therapy
Keywords: Exercise; Physical Activity; Respiratory Failure; Oxygen Inhalation Therapy
MeSH Terms: conditions — Motor Activity; Respiratory Insufficiency | interventions — Surgical Instruments

STUDY DESIGN:
Intervention Model Description: This is a self-controlled study where participants will serve as their own controls. Physical activity levels and quality of life will be measured before and after a 10 week home-based exercise program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Participants (Other): This is a self-controlled study where participants will serve as their own controls. All participants will be enrolled into a 10 week home-based physiotherapy program which will include a total of 2 home visits by a physiotherapist at the start and midpoint of the program. Participants will also receive weekly telephone calls by a research coordinator to provide encouragement for patient on the programme and enquire about compliance to the home exercise regimen and safety (e.g. falls and healthcare utilisation).
  Patients will also be prescribed a lightweight portable oxygen concentrator to facilitate exercise therapy and mobility in the community. They will receive familiarisation and training in its usage as part of the home-based physiotherapy program.
  Interventions: Other: Home-based physiotherapy program; Device: Prescription of a Portable Oxygen Concentrator (POC) device

INTERVENTIONS:
Other: Home-based physiotherapy program — The home-based physiotherapy program will consist of a total of 2 home visits by a physiotherapist which will be scheduled at the start and midpoint of the 10-week program. The visit will include activity education, goal setting and establishment of a home exercise regimen in patient's own home and community environment). Participants will be contacted weekly via telephone to provide encouragement for patient on the program, enquire about compliance to the exercise program and safety (e.g. falls and healthcare utilisation).
Device: Prescription of a Portable Oxygen Concentrator (POC) device — Participants will be prescribed a lightweight Portable Oxygen Concentrator (POC) device [Philips SimplyGo Mini] to be used during exercise and when going into the community setting. Familiarisation and training on the usage of the device will also be provided in conjunction with the home-based physiotherapy program.

SUMMARY:
Long term oxygen therapy (LTOT) is proven to increase the survival of patients with respiratory failure, most commonly from diseases such as Chronic Obstructive Pulmonary Disease (COPD). At least 15 hours' usage per day is needed to improve mortality. Most patients on LTOT utilise bulky oxygen concentrators (OC) which run on continuous Alternating Current (AC) power. This intervention, however, limits patient mobility and social engagement as patients are tethered to their device and confined to their homes.

Reduced physical activity levels have been shown in COPD patients to be associated with reduced quality of life (QoL), increased admission rates to hospital and survival even after adjustment for severity of COPD. Significant benefits stand to be made by improving physical activity levels in LTOT patients. Pulmonary Rehabilitation (PR), which is traditionally conducted in a healthcare setting, is an established intervention that addresses this by improving exercise tolerance but uptake and completion rates have been low due to reasons such as cost and difficulty with transport. LTOT usage is also cited as an independent barrier to PR.

The investigators propose the establishment of a 10-week home-based physiotherapy programme as a novel community-centric and resource-lean intervention that seeks to improve the physical activity level of LTOT patients. Patients will be prescribed an ambulatory oxygen device and receive education on its usage in conjunction with a home exercise regimen which includes a home visit and subsequent telephone support by a physiotherapist in partnership with a community-based healthcare provider.

A prospective pilot study of 30 patients is proposed. The outcome measures include mobility function, activity levels, generic and disease-specific QoL.

If successful, our programme may revolutionize the approach to LTOT patients in Singapore and improve their ability to function independently in the community greatly; in addition, the reduction in hospital-based healthcare utilisation is greatly advantageous.

DETAILED DESCRIPTION:
This will be an investigator-initiated, prospective pilot study which aims to recruit 30 patients in total and conducted over 24 months.

Study Aims and Hypotheses: Utilisation of healthcare resources and burden of care on society for LTOT patients is disproportionately high. The study investigators aim to describe this group of patients and introduce an intervention that aims to promote quality living with a home-based physiotherapy programme.

1. To test the hypothesis that the intervention of a home-based physiotherapy programme together with a lightweight POC will improve physical activity level, reduce daily time spent in sedentary activity, improve Quality of Life (QoL) and reduce symptoms of anxiety and depression of patients on LTOT
2. To describe the functional status of patients on LTOT and their caregivers - physical activity levels, body mass index, psychological, socio-economic background, activities of daily living (ADL) status
3. To describe the barriers to uptake of ambulatory oxygen in patients who fulfil criteria for LTOT
4. As there is a lack of local data on the effectiveness and safety of a home-based physiotherapy program, the study being conducted is a pilot study intended to establish the feasibility of a home-based physiotherapy programme

STUDY BACKGROUND

1. Long-term oxygen therapy (LTOT) is an established medical intervention that has been shown to prolong the survival of a select group of patients with respiratory failure (1, 2). Although local data on the incidence and prevalence of LTOT use in Singapore is lacking, it has been reported in the Danish Oxygen Register that the annual incidence and prevalence of LTOT use in 2010 was 32.2 and 48.1 per 100,000 inhabitants respectively (3). Older studies have reported a LTOT prevalence of 28 per 100,000 in 1992 in the French Oxygen Register (4), LTOT incidence and prevalence of 7.1 and 24 per 100,000 respectively in 2000 in the Swedish Oxygen Register (5) and prevalence of LTOT of 241 per 100,000 in the USA in 1994 (6). Chronic Obstructive Pulmonary Disease (COPD) is by far the main respiratory diagnosis in LTOT patients followed by other diseases such as interstitial lung disease and bronchiectasis (7). In addition, the medical literature has documented rising LTOT usage over the years due to reasons such as increasing survival of COPD patients and increased physician and patient awareness of the benefits of LTOT (8). The costs of LTOT have been recognised to be high, with an estimated 800,000 patients in USA utilising LTOT at cost of approximately $1.4 billion American dollars annually according to a 1995 publication by O'Donohue et al (9). Total Medicare payments for LTOT in 1998 were reported to be USD 1.3 billion (10). A more recent analysis of 329,482 Medicare beneficiaries with COPD who received oxygen from 2001 to 2010 found that 73,659 (22.4%) received oxygen therapy (8).
2. The majority of patients utilise oxygen concentrators (OC) (3,11) which typically run on continuous AC power and weigh between 13-22kg. This intervention, although life-prolonging, nonetheless limits patient mobility as patients are required to utilise oxygen therapy for at least 15 hours a day to benefit. As a result, many patients become confined in their homes.
3. Indeed, patients with chronic respiratory disease requiring LTOT have been reported to be severely limited in their physical activity. Studies of patients on LTOT have shown that 46% of patients walk less than 600m per day (12) and up to 45% are house-bound (13). While this may be due to low exercise tolerance, oxygen therapy may be a contributory factor in itself as patients receiving oxygen from a stationary source often become tethered their device over time. Although there are theoretical benefits to improving exercise tolerance with oxygen therapy (14), it has been reported that patients with severe COPD on LTOT have significantly reduced levels of domestic activity compared with patients with COPD of similar severity but who were not on LTOT (15). Patients with severe COPD and broadly similar health status on LTOT have also been reported to be less independent on activities of daily living than those not requiring LTOT (16).
4. Apart from reduced quality of life, reductions in daily activity levels have been shown to be related to clinically relevant outcomes in COPD patients, such as reduced health status (17), hospital admissions (18, 19) and survival (19) even after adjustment for severity of COPD. Over the years, interest has shifted from improving exercise capacity to increasing daily physical activity (20) which is defined as any bodily movement produced by the contraction of skeletal muscles that increased energy expenditure (21). In fact, it was found in a prospective cohort study of 170 outpatients with stable COPD that objectively measured physical activity was the strongest predictor for all-cause mortality in patients with COPD and that there was a linear association between physical activity and mortality (22). Significant gains in quality of life and reduced utilisation of healthcare stand to be made if the physical activity and mobility profile of patients on LTOT can be increased.
5. An established intervention to improve the mobility and physical activity levels of LTOT patients is Pulmonary Rehabilitation (PR). PR is a structured, multidimensional and multidisciplinary programme over time (at least 6 weeks) that comprises physical training and breathing exercises supervised by a respiratory physiotherapist in conjunction with education guided by objective tests of the respiratory system and exercise capacity such as pulmonary function tests, 6-minute walk test and cardiopulmonary exercise testing. PR been shown to be cost-effective and beneficial in improving shortness of breath, health status and exercise tolerance in patients of all grades of COPD severity, including patients with chronic respiratory failure on LTOT (23).
6. Although the benefits of PR are established, uptake and completion of PR is frequently limited. The percentage of referred participants who did not attend PR at all ranged from 8.3 to 49.6% in a systematic review (24). Many barriers have been cited, such as low referral rates from healthcare providers (25) and low patient and healthcare provider awareness of its availability and benefits. Usage of LTOT has also been found to an independent predictor for non-attendance to PR (26). This is not surprising as patients on LTOT face even greater difficulty than the average patient in participating in PR due to challenges in being able to independently navigate the transportation system to attend outpatient PR whilst on oxygen therapy. Another major barrier worth mentioning is the lack of access from a combination of factors of geography, culture, finances, transportation and other logistics (27, 28). This may be due to the fact that PR is a healthcare-provider centric intervention that is traditionally conducted in a healthcare institution in an outpatient or inpatient setting.
7. Locally in Singapore, patients face a financial disincentive towards participating in PR in the outpatient setting as Medisave, the national medical savings scheme, imposes limits on withdrawals for outpatient healthcare expenditure. Outpatient PR also imposes hidden costs to the patient in the form of transportation and missed days at work for family caregivers who accompany the patient for outpatient PR. Patients are often accompanied by family caregivers or sponsors to healthcare visits in Singapore and the lack of a caregiver to accompany patients for outpatient PR is an important cultural barrier to PR. Inpatient PR in Singapore, on the other hand, is also limited in its capacity to serve many patients due to the national strain on hospital beds. PR clearly has its limitations as a modality in improving the poor physical activity levels of patients on LTOT and a novel solution is needed that addresses the many barriers with PR uptake.
8. The investigators are therefore proposing the establishment of a home-based physiotherapy programme as a novel community and patient-centric and resource-lean intervention that seeks to improve the physical activity of LTOT patients. Patients will be prescribed an ambulatory oxygen device and receive education on its usage in conjunction with a home exercise regimen which would include a home visit by a physiotherapist. It is hypothesised that home-based physiotherapy would be more patient-centric compared to healthcare centre-based physiotherapy as realistic rehabilitation goal settings and exercise regimens can be personalised to each patient's unique home and community environment, lifestyle and care needs. The proposed intervention would be similar to an 8-week home-based PR study recently conducted in the UK which comprised 1 home visit and 7 once-weekly telephone calls from a physiotherapist in the home-based intervention arm which found equivalent short-term outcomes (such as exercise tolerance and dyspnoea-related quality of life) that were equivalent to outpatient centre-based PR (29).
9. Ambulatory Oxygen (AO) is an important enabler in improving the mobility of patients on LTOT in the community and therefore their participation in PR. However there remain many barriers to the uptake of AO such as (i) lack of instruction on the usage of AO, and particularly with regards to AO delivered via oxygen cylinders, (ii) fear of running out of their AO supply while they were using it, (iii) embarrassment and (iv) difficulties with carrying the AO supply (30).
10. These barriers have led to low usage rates of AO via oxygen cylinder with only 39% of patients using AO for more than 2 hours a week in a Danish study published in 1999 (31). In the same study, it was reported that when patients had outdoor activity, the usage of stationary oxygen fell by a couple of hours, resulting in lower overall oxygen usage. This suggested that patients were spending a considerable time outside their home without using their AO (31). In Italy where LTOT is almost exclusively provided by liquid oxygen, it was reported that although most patients (84%) possessed an AO device, only 40% declared that they used it daily with "being ashamed of being seen by passersby with a stroller" being the principal barrier (7). Similar data was presented in a French study which reported that most patients (630/930) used their oxygen only while resting (32).
11. Compared to oxygen cylinders, AO delivered by lightweight Portable Oxygen Concentrator (POC) has the advantages of being (i) user-friendly, (ii) aesthetically more pleasing and is (iii) easily rechargeable with standard household electrical supply (33).

    Such advantages will overcome some of the aforementioned barriers to AO usage.
12. A prospective pilot study of 30 patients is proposed. Assessment of activity levels, QoL and breathlessness will be measured before and after 10 weeks. The 2 components of the proposed intervention, namely the home-based physiotherapy programme and the prescription of a lightweight POC are synergistic in its effects. Supplemental oxygen has been shown to improve exercise duration (34) and therefore rehabilitation while it has been shown that effective use of oxygen was improved by follow-up education, whether given by nurse or physiotherapist, after initiation of oxygen therapy (32). It has been shown that the prescription of AO alone does not automatically assure good adherence to the prescribed treatment or use of AO outdoors (30). The guidance from the home-based physiotherapy programme will comprise of a home visit by a physiotherapist with the aim of reinforcing compliance and usage of AO outside the house, thereby improving the patients' mobility over simply prescribing an AO device. It is hypothesised therefore that patients will be encouraged to use their AO device when they are guided by a home-based physiotherapy programme where rehabilitation goals and exercises are tailored to each patient's unique "life-space" in the home and community.
13. In summary, the proposed intervention of a home-based activity education programme in partnership with a community healthcare provider and in conjunction with a lightweight POC may revolutionize the approach to patients with chronic respiratory failure in Singapore and improve their ability to function independently in the community greatly; in addition, the ability to stay active and community ambulant as well as the reduction the demand on national healthcare resources (e.g. inpatient rehabilitation beds for PR) is greatly advantageous.

Note - References have been cited in subsequent sections

ELIGIBILITY:
Inclusion Criteria (participants are required to fulfill all of the following criteria):

1. Patients aged 21-90 years old who are able to provide informed consent and have their consent signed and dated. Subjects must be able to complete questionnaires.
2. Patients who meet criteria for LTOT i.e. PaO2 ≤55mmHg on room air or PaO2 ≤59mmHg (with pulmonary hypertension, RV hypertrophy, Cor pulmonale, haematocrit ≥55%).
3. Patients should be on LTOT on ≥3 months (to avoid the inclusion of patients who were prescribed oxygen following acute illness).
4. Patients should have clinical stability of their underlying chronic cardiac (e.g. pulmonary hypertension) or respiratory diseases (e.g. COPD, ILD), as demonstrated by no recent acute exacerbation of respiratory/cardiac illness, acute healthcare utilisation (presentation to GP, polyclinic or hospital) or change in medication (or adjustments of non-invasive ventilation) for ≥6 weeks before enrolment.
5. Patients who are sufficiently mobile to perform a 6-minute walk test.

Exclusion Criteria:

1. Patients with any life-threatening condition with a low probability (in the opinion of the investigator) of survival for at least 3 months or who has been hospitalised more than 3 times in the preceding 1 year for respiratory failure.
2. Patients who are not able to ambulate with the lightweight POC (they must be able to perform a 6-minute walk test - this can be unaided or with walking aid) or who have significant limitation of ambulation due to non-respiratory causes such as musculoskeletal (e.g. osteoarthritis) or neuromuscular disease (e.g. Parkinson's disease or stroke), or who are assessed to have no rehabilitation potential.
3. Patients who are actively smoking.
4. Patients who are currently participating in a pulmonary rehabilitation programme.
5. Patients who are pregnant.
6. Patients who are unable or unwilling to complete questionnaires (e.g. patients on LTOT and home mechanical ventilation).

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-09 (Actual); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-03-20 (Estimated)

PRIMARY OUTCOMES:
Change in daily physical activity, which will be measured via the daily step count. | Baseline, 10 weeks
  Daily physical activity will be measured via the daily step count. This will be measured with the activPAL device, a validated tool to measure physical activity. Participants will have the activPAL device applied to their mid-thigh continuously with an adhesive patch for 1 week prior to the home physiotherapy program and for the 10th week of the home physiotherapy program.

SECONDARY OUTCOMES:
Change in respiratory disease specific quality of life questionnaire (St George's Respiratory Questionnaire (SGRQ)) | Baseline, 10 weeks
  Participants will complete the respiratory disease specific quality of life questionnaire St George's Respiratory Questionnaire (SGRQ) at enrollment and after the 10 week home physiotherapy program.
Change in The Hospital Anxiety and Depression Scale (HADS) | Baseline, 10 weeks
  Participants will complete the Hospital Anxiety and Depression Scale (HADS) questionnaire at enrollment and after the 10 week home physiotherapy program to measure the levels of anxiety and depression.
Change in Exercise capacity as measured by 6 minute walk test | Baseline, 10 weeks
  Participants will undergo exercise capacity assessment with the 6-minute walk test .
Change in Exercise capacity assessment with 1 minute Sit to Stand test | Baseline, 10 weeks
  Participants will undergo exercise capacity assessment with the 1-minute Sit to Stand test.
Change in Participants' daily sedentary time | Baseline, 10 weeks
  Daily sedentary time will be measured via the time spent in sedentary body postures (e.g. supine and sitting) as opposed to time spent in active body postures (walking and standing). This will be measured with the activPAL device. Participants will have the activPAL device applied to their mid-thigh continuously for 1 week with an adhesive patch.

CONTACTS AND LOCATIONS:
Overall Officials: Thun How Ong, Dr, Principal Investigator — Department of Respiratory and Critical Care Medicine, Singapore General Hospital
Locations (1):
- Department of Respiratory and Critical Care Medicine, Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Background] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Background] Ringbaek TJ, Lange P. Trends in long-term oxygen therapy for COPD in Denmark from 2001 to 2010. Respir Med. 2014 Mar;108(3):511-6. doi: 10.1016/j.rmed.2013.10.025. Epub 2013 Nov 14. PMID 24275146
- [Background] Chailleux E, Fauroux B, Binet F, Dautzenberg B, Polu JM. Predictors of survival in patients receiving domiciliary oxygen therapy or mechanical ventilation. A 10-year analysis of ANTADIR Observatory. Chest. 1996 Mar;109(3):741-9. doi: 10.1378/chest.109.3.741. PMID 8617085
- [Background] Gustafson T, Lofdahl K, Strom K. A model of quality assessment in patients on long-term oxygen therapy. Respir Med. 2009 Feb;103(2):209-15. doi: 10.1016/j.rmed.2008.09.018. Epub 2008 Nov 5. PMID 18980837
- [Background] Neri M, Melani AS, Miorelli AM, Zanchetta D, Bertocco E, Cinti C, Canessa PA, Sestini P; Educational Study Group of the Italian Association of Hospital Pulmonologists (AIPO). Long-term oxygen therapy in chronic respiratory failure: a Multicenter Italian Study on Oxygen Therapy Adherence (MISOTA). Respir Med. 2006 May;100(5):795-806. doi: 10.1016/j.rmed.2005.09.018. Epub 2005 Oct 20. PMID 16242926
- [Background] Nishi SP, Zhang W, Kuo YF, Sharma G. Oxygen therapy use in older adults with chronic obstructive pulmonary disease. PLoS One. 2015 Mar 18;10(3):e0120684. doi: 10.1371/journal.pone.0120684. eCollection 2015. PMID 25785586
- [Background] O'Donohue WJ Jr, Plummer AL. Magnitude of usage and cost of home oxygen therapy in the United States. Chest. 1995 Feb;107(2):301-2. doi: 10.1378/chest.107.2.301. No abstract available. PMID 7842750
- [Background] Restrick LJ, Paul EA, Braid GM, Cullinan P, Moore-Gillon J, Wedzicha JA. Assessment and follow up of patients prescribed long term oxygen treatment. Thorax. 1993 Jul;48(7):708-13. doi: 10.1136/thx.48.7.708. PMID 8153918
- [Background] Croxton TL, Bailey WC. Long-term oxygen treatment in chronic obstructive pulmonary disease: recommendations for future research: an NHLBI workshop report. Am J Respir Crit Care Med. 2006 Aug 15;174(4):373-8. doi: 10.1164/rccm.200507-1161WS. Epub 2006 Apr 13. PMID 16614349
- [Background] Sandland CJ, Singh SJ, Curcio A, Jones PM, Morgan MD. A profile of daily activity in chronic obstructive pulmonary disease. J Cardiopulm Rehabil. 2005 May-Jun;25(3):181-3. doi: 10.1097/00008483-200505000-00011. PMID 15931024
- [Background] Okubadejo AA, O'Shea L, Jones PW, Wedzicha JA. Home assessment of activities of daily living in patients with severe chronic obstructive pulmonary disease on long-term oxygen therapy. Eur Respir J. 1997 Jul;10(7):1572-5. doi: 10.1183/09031936.97.10071572. PMID 9230249
- [Background] Esteban C, Quintana JM, Aburto M, Moraza J, Egurrola M, Perez-Izquierdo J, Aizpiri S, Aguirre U, Capelastegui A. Impact of changes in physical activity on health-related quality of life among patients with COPD. Eur Respir J. 2010 Aug;36(2):292-300. doi: 10.1183/09031936.00021409. Epub 2010 Jan 14. PMID 20075059
- [Background] Pitta F, Troosters T, Probst VS, Spruit MA, Decramer M, Gosselink R. Physical activity and hospitalization for exacerbation of COPD. Chest. 2006 Mar;129(3):536-44. doi: 10.1378/chest.129.3.536. PMID 16537849
- [Background] Garcia-Aymerich J, Lange P, Benet M, Schnohr P, Anto JM. Regular physical activity reduces hospital admission and mortality in chronic obstructive pulmonary disease: a population based cohort study. Thorax. 2006 Sep;61(9):772-8. doi: 10.1136/thx.2006.060145. Epub 2006 May 31. PMID 16738033
- [Background] Wouters EFM, Franssen FME, Spruit MA. Survival and physical activity in COPD: a giant leap forward! Chest. 2011 Aug;140(2):279-281. doi: 10.1378/chest.11-0521. No abstract available. PMID 21813522
- [Background] Waschki B, Kirsten A, Holz O, Muller KC, Meyer T, Watz H, Magnussen H. Physical activity is the strongest predictor of all-cause mortality in patients with COPD: a prospective cohort study. Chest. 2011 Aug;140(2):331-342. doi: 10.1378/chest.10-2521. Epub 2011 Jan 27. PMID 21273294
- [Background] Carone M, Patessio A, Ambrosino N, Baiardi P, Balbi B, Balzano G, Cuomo V, Donner CF, Fracchia C, Nava S, Neri M, Pozzi E, Vitacca M, Spanevello A. Efficacy of pulmonary rehabilitation in chronic respiratory failure (CRF) due to chronic obstructive pulmonary disease (COPD): The Maugeri Study. Respir Med. 2007 Dec;101(12):2447-53. doi: 10.1016/j.rmed.2007.07.016. Epub 2007 Aug 28. PMID 17728121
- [Background] Keating A, Lee A, Holland AE. What prevents people with chronic obstructive pulmonary disease from attending pulmonary rehabilitation? A systematic review. Chron Respir Dis. 2011;8(2):89-99. doi: 10.1177/1479972310393756. PMID 21596892
- [Background] Jones SE, Green SA, Clark AL, Dickson MJ, Nolan AM, Moloney C, Kon SS, Kamal F, Godden J, Howe C, Bell D, Fleming S, Haselden BM, Man WD. Pulmonary rehabilitation following hospitalisation for acute exacerbation of COPD: referrals, uptake and adherence. Thorax. 2014 Feb;69(2):181-2. doi: 10.1136/thoraxjnl-2013-204227. Epub 2013 Aug 14. PMID 23945168
- [Background] Hayton C, Clark A, Olive S, Browne P, Galey P, Knights E, Staunton L, Jones A, Coombes E, Wilson AM. Barriers to pulmonary rehabilitation: characteristics that predict patient attendance and adherence. Respir Med. 2013 Mar;107(3):401-7. doi: 10.1016/j.rmed.2012.11.016. Epub 2012 Dec 19. PMID 23261311
- [Background] Thorpe O, Kumar S, Johnston K. Barriers to and enablers of physical activity in patients with COPD following a hospital admission: a qualitative study. Int J Chron Obstruct Pulmon Dis. 2014 Jan 21;9:115-28. doi: 10.2147/COPD.S54457. eCollection 2014. PMID 24489465
- [Background] Holland AE, Mahal A, Hill CJ, Lee AL, Burge AT, Cox NS, Moore R, Nicolson C, O'Halloran P, Lahham A, Gillies R, McDonald CF. Home-based rehabilitation for COPD using minimal resources: a randomised, controlled equivalence trial. Thorax. 2017 Jan;72(1):57-65. doi: 10.1136/thoraxjnl-2016-208514. Epub 2016 Sep 26. PMID 27672116
- [Background] Arnold E, Bruton A, Donovan-Hall M, Fenwick A, Dibb B, Walker E. Ambulatory oxygen: why do COPD patients not use their portable systems as prescribed? A qualitative study. BMC Pulm Med. 2011 Feb 11;11:9. doi: 10.1186/1471-2466-11-9. PMID 21314932
- [Background] Ringbaek T, Lange P, Viskum K. Compliance with LTOT and consumption of mobile oxygen. Respir Med. 1999 May;93(5):333-7. doi: 10.1016/s0954-6111(99)90314-1. PMID 10464899
- [Background] Pepin JL, Barjhoux CE, Deschaux C, Brambilla C. Long-term oxygen therapy at home. Compliance with medical prescription and effective use of therapy. ANTADIR Working Group on Oxygen Therapy. Association Nationale de Traitement a Domicile des Insuffisants Respiratories. Chest. 1996 May;109(5):1144-50. doi: 10.1378/chest.109.5.1144. PMID 8625658
- [Background] Dunne PJ. The clinical impact of new long-term oxygen therapy technology. Respir Care. 2009 Aug;54(8):1100-11. PMID 19650950
- [Background] Voduc N, Tessier C, Sabri E, Fergusson D, Lavallee L, Aaron SD. Effects of oxygen on exercise duration in chronic obstructive pulmonary disease patients before and after pulmonary rehabilitation. Can Respir J. 2010 Jan-Feb;17(1):e14-9. doi: 10.1155/2010/142031. PMID 20186361